CLINICAL TRIAL: NCT01768273
Title: A Phase 1, Open-label, Multi-Dose Study to Assess Pharmacokinetic Interaction Between PA-824 and Midazolam
Brief Title: Evaluation of the Pharmacokinetic Interaction Between PA-824 and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-824-CL-006
Record Dates: First submitted 2013-01-07; First posted 2013-01-15 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
Keywords: PA-824,; midazolam; drug-drug interaction; pharmacokinetics; pretomanid; CL-006
MeSH Terms: conditions — Tuberculosis | interventions — Midazolam; pretomanid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam and 824 (Experimental): 2 mg midazolam (oral syrup) Day 1 and Day 17. 400 mg PA-824 once daily Day 4 - 17.
  Interventions: Drug: Midazolam; Drug: PA-824

INTERVENTIONS:
Drug: Midazolam
  Other Names: Dormicum; Hypnovel; Versed
Drug: PA-824

SUMMARY:
The purpose of this study is to determine the safety and tolerability of PA-824 when given with a single dose of midazolam, and to determine whether PA-824 inhibits CYP3A to a clinically important degree as measured by the effect of PA-824 on the pharmacokinetics of midazolam, a known CYP3A substrate.

DETAILED DESCRIPTION:
This study is an open-label, fixed sequence design. 14 subjects will receive a single dose of 2 mg midazolam, followed by a 2-day wash-out. Following the wash-out, all subjects will receive PA-824 once daily for 14 days. All patients will receive a single dose of 2 mg midazolam on the 14th day of PA-824 dosing. This study will evaluate 400 mg PA-824.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, have provided written informed consent (as evidenced by signature on an informed consent document approved by an IRB), and agree to abide by the study restrictions.
2. Be healthy non-tobacco/nicotine using (6-month minimum) adult subjects, 19 to 50 years of age, inclusive.
3. Be medically healthy subjects with clinically insignificant Screening results (among laboratory profiles, medical histories, ECGs, or physical exam), as deemed by the Principal Investigator.
4. Have a body mass index of 18 to 29.
5. Have negative urine test results for alcohol and drugs of abuse such as amphetamines, cannabinoids, and cocaine metabolites at both Screening and Check-in.
6. Agree to follow the requirements set forth in the protocol regarding pregnancy controls and donation of sperm, blood, or blood components.

Exclusion Criteria:

Medical History

1. Any clinically significant (as deemed by the Principal Investigator) history, acute illness (resolved within 4 weeks of screening), or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic, psychological, or psychiatric disease.
2. History of peptic ulcer disease, gastritis, esophagitis, or gastroesophageal reflux disease.
3. History of any clinically significant cardiac abnormality (as deemed by the Principal Investigator).
4. Any clinically significant ECG abnormality at Screening (as deemed by the Principal Investigator and the Sponsor's Medical Monitor)

   Note: the following can be considered not clinically significant without consulting Sponsor's Medical Monitor:
   * Heart rate ≥50 beats per minute (sinus bradycardia with heart rate between 45 and 49, inclusive, is acceptable only in younger athletic subjects)
   * Mild first degree A-V block (P-R interval <0.23 sec)
   * Right or left axis deviation
   * Incomplete right bundle branch block
   * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
5. History of prolonged QT interval.
6. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease or CHF or terminal cancer)
7. Resting pulse rate < 40 or > 100 bpm at Screening.
8. At Screening blood pressure greater than 140/90 mm Hg or below 95/65 mm Hg (supine, after a minimum 5-minute supine rest)
9. At either Screening or the pre-dose read before the first dose, a QTcB (Bazett's correction) >450ms for men and women, calculated from the average of triplicate reads collected at the screening and predose sitting.
10. At either Screening or the pre-dose read before the first dose, a QTcF (Fridericia's correction) >450ms for men and women, calculated from the average of triplicate reads collected at the screening and predose sitting.
11. History of hypokalemia or hypomagnesemia.
12. History or presence of alcoholism or drug abuse within the past 2 years (as deemed by the Principal Investigator).
13. Use of alcohol within 72 hours prior to dosing.
14. Significant history of drug and/or food allergies (as deemed by the Principal Investigator).
15. For women, subject is pregnant (positive test for serum HCG at Screening or Check-in), breastfeeding or planning to conceive a child within 30 days of cessation of treatment.
16. For males, planning to father a child within 12 weeks of cessation of treatment.
17. History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination.

    Specific Treatments
18. Any contraindication to the use of nitroimidazoles, or prior treatment with PA-824 or OPC-67683.
19. Use of any systemic or topical prescription medication within 14 days prior to dosing or during the study, except hormonal contraceptives in women.
20. Use of any systemic or over-the-counter medication including vitamins, herbal preparations, antacids, cough and cold remedies, etc., within 7 days prior to dosing or during the study treatment periods.
21. Use of any drugs or substances within 30 days prior to dosing, known to be strong inhibitors or inducers of cytochrome P450 enzymes (including quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan, etc.) or known to prolong the QT interval (including amiodarone, bepridil chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, quinolones, sotalol, sparfloxacin, thioridazine,) or barbiturates, opiates, or phenothiazines.
22. Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine, etc.) within 30 days prior to dosing.
23. Consumption of products containing grapefruit within 10 days prior to dosing.
24. Any special dietary changes during the 30 days prior to dosing, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
25. Any strenuous exercise within 7 days of Check-in, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
26. Donation of whole blood or significant loss of blood within 56 days prior to dosing.
27. Plasma donation within 7 days prior to dosing.
28. Participation in another interventional clinical trial within 30 days prior to dosing.

    Based on Lab Abnormalities
29. Any serum creatinine or BUN measure beyond the upper limit of the normal range at Screening or Check-in. Individual values may be discussed with the Sponsor Medical Monitor.
30. Hemoglobin < 12.0 g/dL at the screening visit.
31. Positive Screening test for HCV, HBV, or HIV.
32. Any other factor which suggests to the Principal Investigator that the subject should not participate in the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of multiple-dose administration of PA-824 on the pharmacokinetics of midazolam, a sensitive probe substrate and representative compound for drugs metabolized by CYP3A enzymes. | Day 18
  The PK parameters to be calculated for midazolam and 1-hydroxy midazolam include area under the curve [AUC(0-t) and AUC(0-inf)], maximum observed concentration (Cmax), time to maximum observed plasma concentration (Tmax), half-life (t1/2), and apparent terminal elimination rate constant (Kel).
To evaluate the safety and tolerability of PA-824 when given with midazolam. | Day 108
  Safety assessments include clinical laboratory assessments, vital signs including respiration rates, electrocardiograms (ECGs), physical examinations, ophthalmology examinations, including visual acuity tests and slit lamp examinations, and monitoring of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- See also: Related Info — http://www.tballiance.org